CLINICAL TRIAL: NCT01008137
Title: Cell-mediated Immunity Study of H1N1 Influenza A Vaccine With Trivalent Inactivated Influenza Vaccine in Healthy Adults
Brief Title: Sinovac, H1N1 Vaccine + Trivalent Inactivated Influenza Vaccine, Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO-PanFlu-4002
Record Dates: First submitted 2009-10-29; First posted 2009-11-05 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Care Provider

ARMS (3):
- Group 1: Day 0-PANFLU.1; Day 21-ANFLU (Experimental): 50 subjects to receive-Day 0: 15 μg PANFLU.1 vaccine; Day 21: 15 μg ANFLU vaccine.
  Interventions: Biological: H1N1 influenza A Vaccine (PANFLU.1); Biological: Trivalent Inactivated Influenza Vaccine (ANFLU)
- Group 2: Day 0-ANFLU; Day 21-PANFLU.1 (Experimental): 50 subjects to receive-Day 0: 15 μg ANFLU vaccine; Day 21: 15 μg PANFLU.1 vaccine.
  Interventions: Biological: H1N1 influenza A Vaccine (PANFLU.1); Biological: Trivalent Inactivated Influenza Vaccine (ANFLU)
- Group 3: Day 0-PANFLU.1+ANFLU (Experimental): 50 subjects to receive-Day 0: 15 μg PANFLU.1 vaccine+ANFLU vaccine.
  Interventions: Biological: H1N1 influenza A Vaccine (PANFLU.1); Biological: Trivalent Inactivated Influenza Vaccine (ANFLU)

INTERVENTIONS:
Biological: H1N1 influenza A Vaccine (PANFLU.1) — H1N1 influenza A Vaccine (PANFLU.1), 15 micrograms per dose. Vaccines will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm (randomized in one arm)
Biological: Trivalent Inactivated Influenza Vaccine (ANFLU) — Trivalent Inactivated Influenza Vaccine (ANFLU), 15 micrograms per dose. Vaccines will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm (injected in the other arm)

SUMMARY:
A single center, randomized clinical trial is to be conducted in healthy adults (18-60 years) to evaluate the safety and immunogenicity and study the cell-mediated Immunity of Sinovac's H1N1 influenza A Vaccine (PANFLU.1) with Trivalent Inactivated Influenza Vaccine (ANFLU).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged between 18 and 60
2. Be able to show legal identity card for the sake of recruitment
3. Volunteers are able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. History of H1N1 vaccine or seasonal influenza vaccine administration
3. Women of pregnancy, lactation or about to be pregnant in 60 days
4. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
5. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
6. Autoimmune disease or immunodeficiency
7. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
8. Diabetes mellitus (type I or II), with the exception of gestational diabetes
9. History of thyroidectomy or thyroid disease that required medication within the past 12 months
10. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
11. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
12. Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
13. Seizure disorder other than:

    * Febrile seizures under the age of two years old
    * Seizures secondary to alcohol withdrawal more than 3 years ago, or
    * A singular seizure not requiring treatment within the last 3 years
14. Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
15. Guillain-Barre Syndrome
16. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
17. History of any blood products within 3 months before the dosing
18. Administration of any other investigational research agents within 30 days before the dosing
19. Administration of any live attenuated vaccine within 30 days before the dosing
20. Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
21. Be receiving anti-TB prophylaxis or therapy currently
22. Axillary temperature > 37.0 centigrade at the time of dosing
23. Psychiatric condition that precludes compliance with the protocol:

    * Past or present psychoses
    * Past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years
    * Disorder requiring lithium
    * Suicidal ideation occurring within five years prior to enrollment
24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Study the cell-mediated immunity of H1N1 vaccine with seasonal influenza vaccine | 6 months

SECONDARY OUTCOMES:
Evaluate immunogenicity of H1N1 vaccine with seasonal influenza vaccine in adults | 3 months
Evaluate safety of H1N1 vaccine with seasonal influenza vaccine in adults | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Centers for Diseases Control and Prevention, Beijing, China

REFERENCES:
- [Derived] Wu J, Zhong X, Li CK, Zhou JF, Lu M, Huang KY, Dong M, Liu Y, Luo FJ, Du N, Chui C, Liu LQ, Smith NM, Li B, Shi NM, Song LF, Gao Y, Wang DY, Wang X, Zhu WF, Yan Y, Li Z, Chen JT, McMichael AJ, Yin WD, Xu XN, Shu Y. Optimal vaccination strategies for 2009 pandemic H1N1 and seasonal influenza vaccines in humans. Vaccine. 2011 Jan 29;29(5):1009-16. doi: 10.1016/j.vaccine.2010.11.058. Epub 2010 Dec 2. PMID 21130194